CLINICAL TRIAL: NCT06931977
Title: Wellness and Epigenetic Impact of a Natural Product Supplement System Combined With Lifestyle Modification
Brief Title: Natural Product System and Lifestyle Modification
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: dōTERRA International (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: DO-125023-FWS
Record Dates: First submitted 2025-04-02; First posted 2025-04-17 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Healthy
Keywords: Gene expression; Essential oil; Copaiba; Omega 3; Probiotic; Greens powder

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Participants and investigators will be masked to whether the participants receive the copaiba essential oil or placebo, but will know the identity of the other three supplements they take.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supplement System + Copaiba softgels (Experimental): Participants in this arm will take one VMG sachet, three EOM softgels, and one copaiba softgel in the morning with food. At least eight hours later, they will take one PBR capsule and one copabia softgel with food. They will follow this dosing regimen every day for 12 weeks.
  Interventions: Dietary Supplement: Supplement system + copaiba softgels
- Supplement System + placebo softgels (Placebo Comparator): Participants in this arm will take one VMG sachet, three EOM softgels, and one placebo softgel in the morning with food. At least eight hours later, they will take one PBR capsule and one placebo softgel with food. They will follow this dosing regimen every day for 12 weeks.
  Interventions: Dietary Supplement: Supplement system + placebo softgels

INTERVENTIONS:
Dietary Supplement: Supplement system + copaiba softgels — The supplement system consists of:
  * dōTERRA VMG+ Whole-Food Nutrient Complex (VMG) sachets
  * dōTERRA EO Mega+ Essential Oil Omega Complex (EOM) softgels
  * dōTERRA PB Restore ProBiome Complex (PBR) capsules
  Which will also be taken with:
  • dōTERRA Copaiba Essential Oil (CEO) softgels
  VMG is a powdered nutritional drink packaged in individual sachets. The powder is a blend of food powders/extracts, vitamins and minerals, probiotics, essential oils, and sweeteners.
  EOM is a softgel containing fish oil and wild orange essential oil.
  PBR is a capsule containing a mix of pre-, pro-, and post-biotics and bacteriophages.
  CEO is a softgel containing Copaifera (copaiba) essential oil and extra virgin olive oil.
  Participants will also be asked to implement lifestyle changes. They will be asked to try to get at least 8 hours of sleep, eat at least three servings of fruit/vegetables daily, and exercise at least 30 minutes every day.
  Arms: Supplement System + Copaiba softgels
Dietary Supplement: Supplement system + placebo softgels — The supplement system consists of:
  * dōTERRA VMG+ Whole-Food Nutrient Complex (VMG) sachets
  * dōTERRA EO Mega+ Essential Oil Omega Complex (EOM) softgels
  * dōTERRA PB Restore ProBiome Complex (PBR) capsules
  Which will also be taken with:
  • Olive oil placebo softgels
  VMG is a powdered nutritional drink packaged in individual sachets. The powder is a blend of food powders/extracts, vitamins and minerals, probiotics, essential oils, and sweeteners.
  EOM is a softgel containing fish oil and wild orange essential oil.
  PBR is a capsule containing a mix of pre-, pro-, and post-biotics and bacteriophages.
  The placebo is a softgel containing extra virgin olive oil.
  Participants will also be asked to implement lifestyle changes. They will be asked to try to get at least 8 hours of sleep, eat at least three servings of fruit/vegetables daily, and exercise at least 30 minutes every day.
  Arms: Supplement System + placebo softgels

SUMMARY:
The goal of this clinical trial is to learn whether four dietary supplements and lifestyle changes can affect gene expression and blood markers in healthy volunteers. The main questions it aims to answer are:

1. How does daily ingestion of dietary supplements affect gene expression and hsCRP and vitamin D levels measured in blood?
2. How does daily ingestion of dietary supplements affect anthropometric measurements, sleep and physical activity, and gut microbiome composition?
3. How does daily ingestion of dietary supplements affect cognitive and subjective health parameters?
4. Do prescriptive lifestyle modifications affect the supplements' efficacy?
5. Is there a difference in outcomes between participants who take all four study supplements and those who take three study supplements with a placebo?
6. Is ingesting dietary supplements for 12 weeks safe, as measured by laboratory tests and adverse events?

DETAILED DESCRIPTION:
This double-blind, repeated measures study will recruit healthy adults to determine efficacy, safety, anthropometric, microbiome, and epigenetic effects of consuming four dietary supplements daily for 12 weeks. Prescriptive lifestyle modifications (diet, exercise, and sleep) will be evaluated with the supplement use.

ELIGIBILITY:
Inclusion Criteria:

* Adults ages 30-55 years old
* Willing to attend three study visits at Prime Meridian Health Clinic in Pleasant Grove, Utah
* Willing and able to undergo three blood draws over 12 weeks
* Willing to provide urine and stool samples three times over 12 weeks
* Willing to wash out of all internally consumed essential oils or botanical products for at least 2 weeks prior to starting the study, and willing to maintain the washout for the duration of the study (14 weeks).
* Willing to wash out of all fish oil supplements, probiotic supplements, and greens powder mix 2 weeks prior to starting the study, and willing to maintain the washout for the duration of the study (14 weeks).
* Willing and able to consume study product as directed daily for about 12 weeks
* Willing to track consumption of study product
* Willing to implement changes to diet, exercise, and sleep habits for 12 weeks
* Willing to avoid alcohol, recreational drugs, and smoking/vaping for the duration of the study (approximately 12 weeks)
* Own a smartphone or tablet and willing to download the fitness tracker app
* Willing to wear a fitness tracker for the duration of the study (approximately 12 weeks)
* At least 110 pounds
* No metabolic disease (BMI>35, diagnosis and treatment of
* hypertension, diabetes, or dyslipidemia)
* No major diseases under treatment by doctor (Medical Reviewer's
* discretion)
* No pregnancy within the last 60 days or currently breastfeeding
* (females)
* No allergy to any of the ingredients in the study products
* No regular internal consumption of the study products within the last 1 month (regularly is defined as dosing daily for more than 2 consecutive weeks, or dosing more than 2-3 times per week for 4 consecutive weeks)
* No alcohol, recreational drug, or smoking/vaping use in the past 1 month
* No evidence of medical condition, significant disease or disorder, medication, or surgery within the past 12 months that may, in the judgment of the medical provider, put the participant at risk or affect study results, procedures, or outcomes
* Not currently or previously participating in any other clinical trial within the last 30 calendar days

Exclusion Criteria:

* Failure to meet all listed inclusion criteria

Ages: 30 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 120 (Estimated)
Dates: Start 2025-04-29 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Gene expression | 12 weeks
  Gene expression analysis refers to a genome-wide quantification of methylation. EPIC850k array will be used for methylation analysis. This represents approximately 900,000 gene locations. The main feature performed is a differential methylation analysis to determine what has significantly changed from one time point to another.
Vitamin D 25-hydroxy (ng/mL) | 12 weeks
  Serum marker for Vitamin D levels
High sensitivity C-reactive protein (mg/L) | 12 weeks
  Serum marker for hsCRP levels

SECONDARY OUTCOMES:
Albumin (g/dL) | 12 weeks
  Item in comprehensive metabolic panel for safety assessment
Blood urea nitrogen (BUN) (mg/dL) | 12 weeks
  Item in comprehensive metabolic panel for safety assessment
Creatinine (mg/dL) | 12 weeks
  Item in comprehensive metabolic panel for safety assessment
Alkaline phosphatase (U/L) | 12 weeks
  Item in comprehensive metabolic panel for safety assessment
Alanine transaminase (ALT) (U/L) | 12 weeks
  Item in comprehensive metabolic panel for safety assessment
Aspartate aminotransferase (AST) (U/L) | 12 weeks
  Item in comprehensive metabolic panel for safety assessment
Calcium (mg/dL) | 12 weeks
  Item in comprehensive metabolic panel for safety assessment
Carbon Dioxide (mmol/L) | 12 weeks
  Item in comprehensive metabolic panel for safety assessment
Chloride (mmol/L) | 12 weeks
  Item in comprehensive metabolic panel for safety assessment
Potassium (mmol/L) | 12 weeks
  Item in comprehensive metabolic panel for safety assessment
Sodium (mmol/L) | 12 weeks
  Item in comprehensive metabolic panel for safety assessment
Total bilirubin (mg/dL) | 12 weeks
  Item in comprehensive metabolic panel for safety assessment
Total protein (g/dL) | 12 weeks
  Item in comprehensive metabolic panel for safety assessment
White blood cells (x10E3/uL) | 12 weeks
  Item in complete blood count for safety assessment
Red blood cells (x10E6/uL) | 12 weeks
  Item in complete blood count for safety assessment
Hemoglobin (g/dL) | 12 weeks
  Item in complete blood count for safety assessment
Hematocrit (%) | 12 weeks
  Item in complete blood count for safety assessment
Mean corpuscular volume (fL) | 12 weeks
  Item in complete blood count for safety assessment
Mean corpuscular hemoglobin concentration (g/dL) | 12 weeks
  Item in complete blood count for safety assessment
Red cell distribution width (%) | 12 weeks
  Item in complete blood count for safety assessment
Platelets (x10E3/uL) | 12 weeks
  Item in complete blood count for safety assessment
Neutrophils (%) | 12 weeks
  Item in complete blood count for safety assessment
Monocytes (%) | 12 weeks
  Item in complete blood count for safety assessment
Eosinophils (%) | 12 weeks
  Item in complete blood count for safety assessment
Basophils (%) | 12 weeks
  Item in complete blood count for safety assessment
Neutrophils (Absolute) (x10E3/uL) | 12 weeks
  Item in complete blood count for safety assessment
Lymphocytes (Absolute) (x10E3/uL) | 12 weeks
  Item in complete blood count for safety assessment
Monocytes (Absolute) (x10E3/uL) | 12 weeks
  Item in complete blood count for safety assessment
Eosinophils (Absolute) (x10E3/uL) | 12 weeks
  Item in complete blood count for safety assessment
Basophils (Absolute) (x10E3/uL) | 12 weeks
  Item in complete blood count for safety assessment
Immature granulocytes (%) | 12 weeks
  Item in complete blood count for safety assessment
Immature granulocytes (Absolute) (x10E3/uL) | 12 weeks
  Item in complete blood count for safety assessment
Adverse events | 12 weeks
  This study will monitor the occurrence and frequency of adverse events and safety, both through participant report and blood chemistry/hematology/urine analyses.
Generalized Anxiety Disorder-7 (GAD-7) scale | 12 weeks
  Validated, self-reported scale for the measurement of anxiety severity. The GAD-7 is a 7-item scale with total scores between 0 and 21. Higher scores indicate higher anxiety severity.
Patient Health Questionnaire (PHQ-8) scale | 12 weeks
  Validated, self-reported scale for the measurement of depression severity. The PHQ-8 is an 8-item scale with total scores between 0 and 12. Higher scores indicate higher depression severity.
Leeds Sleep Evaluation Questionnaire (LSEQ) scale | 12 weeks
  Validated, self-reported scale for the measurement of sleep quality. The LSEQ is a 10-item scale. Each item is scored 0 to 100. Higher scores indicate better sleep quality.
Short Form-20 (SF-20) scale | 12 weeks
  Validated, self-reported scale for the assessment of subjective quality of life. The SF-20 is a 20-item scale. Each item is scored 0-100. Higher scores indicate better subjective quality of life.
Digestion-associated Quality of Life Questionnaire (DQLQ) | 12 weeks
  Validated, self-reported scale for the measurement of digestion-associated quality of life outcomes. The DQLQ is a 9-item scale with total scores between 0 and 9. Each item is scored as a percentage 0-100, with 100 representing a score of 1. Higher scores indicate greater dissatisfaction with digestion-associated quality of life outcomes.
Gastrointestinal Symptom Rating Scale (GSRS) | 12 weeks
  Validated, self-reported scale for the assessment of gastrointestinal symptoms and how much discomfort they cause. The GSRS consists of 15 items scored between 1 and 7 each. Higher scores indicate more severe symptoms.
Digit Symbol Substitution Test (DSST) | 12 weeks
  A timed test that measures psychomotor performance and cognitive function. The test taker is given a key grid of numbers and matching symbols, and a list of numbers and empty boxes. The test taker matches the symbols to the numbers in the empty boxes within the allowed time (90 seconds). Participants will be scored according to the number of symbols they correctly correlate with a number.
Word Recall Test (WRT) | 12 weeks
  A timed memory assessment that asks the test taker to recall a list of words. The test administrator reads a list of 15 words, and the test taker is asked to immediately write down all the words they remember. After 15 minutes, the test taker is asked to write down the words again. Participants will be scored based on the number of words they recall immediately and after 15 minutes.
Functional movement test | 12 weeks
  Functional Movement Test (FMT) is an assessment used to evaluate an individual's movement patterns, mobility, stability, and overall functional fitness. It consists of several fundamental movement tests designed to identify weaknesses, imbalances, or limitations in a person's functional ability. During an FMT, a person is asked to perform movements such as directional neck movements, arm reaches, squats, push-ups, and balance on one leg. Each movement is scored based on form and control.
Gut microbiome test | 12 weeks
  Participants complete stool collection kits. Stool is analyzed for gut microbiome composition (e.g. bacteria %/count/type)
Total steps | 12 weeks
  Daily number of steps measured with fitness trackers.
Sleep score | 12 weeks
  A personalized score, ranging from 1 to 100, that reflects quality of sleep based on factors like time asleep, deep and REM sleep.
Body mass index (BMI) | 12 weeks
  A calculation of body fat based on height and weight
Body mass percentage (%) | 12 weeks
  An estimation of bone, fat, muscle, and water mass %
Blood pressure (mmHg) | 12 weeks
  The force of blood pushing against the walls of arteries.
Heart rate (BPM) | 12 weeks
  The number of heart beats per minute
Waist circumference (cm) | 12 weeks
  The circumference of the waist measured at the thinnest point of the waist
Insulin (uIU/mL) | 12 weeks
  Serum marker used to determine insulin levels
Sex hormone binding globulin (nmol/L) | 12 weeks
  Serum marker used to determine SHBG (Sex Hormone Binding Globulin) levels
Testosterone (ng/dL) | 12 weeks
  Serum marker used to determine testosterone levels
Thyroxine (T4) (ng/dL) | 12 weeks
  Serum marker used to determine thyroxine (T4) levels
Thyroglobulin antibody (IU/mL) | 12 weeks
  Serum marker used to determine thyroglobulin antibody levels
Thyroid peroxidase antibody (IU/mL) | 12 weeks
  Serum marker used to determine thyroid peroxidase antibody levels
Vitamin B12 (pg/mL) | 12 weeks
  Serum marker used to determine Vitamin B12 levels
Ferritin (ng/mL) | 12 weeks
  Serum marker used to determine ferritin levels
Gamma-glutamyl transferase (GGT) | 12 weeks
  Serum marker used to determine GGT levels
Transferritin saturation | 12 weeks
  Serum test used to determine UIBC, TIBC, Iron, Fe Saturation%
Total sleep (minutes) | 12 weeks
  Total number of minutes asleep, as measured by fitness tracker.
Light sleep (%) | 12 weeks
  The percentage of time asleep spent in light sleep, as measured by fitness tracker.
Deep sleep (%) | 12 weeks
  The percentage of time asleep spent in deep sleep, as measured by fitness tracker.
REM sleep (%) | 12 weeks
  The percentage of time asleep spent in deep sleep, as measured by fitness tracker.
Active minutes | 12 weeks
  Number of daily active minutes as measured by fitness tracker.
Sedentary minutes | 12 weeks
  Number of daily sedentary minutes as measured by fitness tracker.
Active calories burned | 12 weeks
  Number of daily active calories burned as measured by fitness tracker.
Total calories burned | 12 weeks
  Number of daily total calories burned as measured by fitness tracker.

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Stevens, PhD, Principal Investigator — doTERRA International LLC
Locations (1):
- doTERRA International, Pleasant Grove, Utah, United States

IPD SHARING:
Plan to Share IPD: No